CLINICAL TRIAL: NCT02847026
Title: Immunogenicity of a Booster Dose of Fractional Inactivated Poliovirus Vaccine (fIPV) Delivered Intradermally Concomitantly With Rotavirus Vaccines
Brief Title: Fractional Inactivated Poliovirus Vaccine Booster and Rotavirus Study
Acronym: fIPV
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ICDDRB-RRC-PR-15105
Record Dates: First submitted 2016-07-25; First posted 2016-07-27 (Estimated); Last update posted 2018-07-18 (Actual); Status verified 2016-08

CONDITIONS: Poliomyelitis
Keywords: inactivated poliovirus vaccine; fractional inactivated poliovirus vaccine; Rotavirus; Rotarix; RotaTeq; fIPV; IPV
MeSH Terms: conditions — Poliomyelitis | interventions — Aging; RIX4414 vaccine; RotaTeq

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- IPV at 14 and 22 weeks of age, Rotarix (Active Comparator): Participants in this arm will receive a full dose of IPV at 14 weeks of age and a full dose IPV booster at 22 weeks of age. Rotarix will also be given at 6 and 10 weeks of age.
  Interventions: Biological: IPV at 14 and 22 weeks of age, Rotarix
- IPV at 14 and 22 weeks of age, RotaTeq (Active Comparator): Participants in this arm will receive a full dose of IPV at 14 weeks of age and a full dose IPV booster at 22 weeks of age. RotaTeq will also be given at 6, 10, and 14 weeks of age.
  Interventions: Biological: IPV at 14 and 22 weeks of age, RotaTeq
- IPV at 14 and fIPV at 22 weeks, Rotarix (Active Comparator): Participants in this arm will receive a full dose of IPV at 14 weeks of age and a fractional dose IPV (fIPV) booster at 22 weeks of age. Rotarix will also be given at 6 and 10 weeks of age.
  Interventions: Biological: IPV at 14 and fIPV at 22 weeks, Rotarix
- IPV at 14 and fIPV at 22 weeks, RotaTeq (Active Comparator): Participants in this arm will receive a full dose of IPV at 14 weeks of age and a fractional dose IPV (fIPV) booster at 22 weeks of age. RotaTeq will also be given at 6, 10, and 14 weeks of age.
  Interventions: Biological: IPV at 14 and fIPV at 22 weeks, RotaTeq
- IPV at 6 and fIPV at 22 weeks, Rotarix (Active Comparator): Participants in this arm will receive a full dose of IPV at 6 weeks of age and a fractional dose IPV (fIPV) booster at 22 weeks of age. Rotarix will also be given at 6 and 10 weeks of age.
  Interventions: Biological: IPV at 6 and fIPV at 22 weeks, Rotarix
- IPV at 6 and fIPV at 22 weeks, RotaTeq (Active Comparator): Participants in this arm will receive a full dose of IPV at 6 weeks of age and a fractional dose IPV (fIPV) booster at 22 weeks of age. RotaTeq will also be given at 6, 10, and 14 weeks of age.
  Interventions: Biological: IPV at 6 and fIPV at 22 weeks, RotaTeq
- fIPV at 6-14-22 weeks of age, Rotarix (Active Comparator): Participants in this arm will receive fractional doses of IPV (fIPV) at 6 and 14 weeks of age and a fIPV booster at 22 weeks of age. Rotarix will also be given at 6 and 10 weeks of age.
  Interventions: Biological: fIPV at 6-14-22 weeks of age, Rotarix
- fIPV at 6-14-22 weeks of age, RotaTeq (Active Comparator): Participants in this arm will receive fractional doses of IPV (fIPV) at 6 and 14 weeks of age and a fIPV booster at 22 weeks of age. RotaTeq will also be given at 6, 10, and 14 weeks of age.
  Interventions: Biological: fIPV at 6-14-22 weeks of age, RotaTeq

INTERVENTIONS:
Biological: IPV at 14 and 22 weeks of age, Rotarix — Participants in this arm will receive a full dose of inactivated poliovirus vaccine (IPV) at 14 weeks of age and a full dose IPV booster at 22 weeks of age. They will also receive the rotavirus vaccine, Rotarix, at 6 and 10 weeks of age.
  Arms: IPV at 14 and 22 weeks of age, Rotarix
Biological: IPV at 14 and 22 weeks of age, RotaTeq — Participants in this arm will receive a full dose of inactivated poliovirus vaccine (IPV) at 14 weeks of age and a full dose IPV booster at 22 weeks of age. They will also receive the rotavirus vaccine, RotaTeq, at 6, 10, and 14 weeks of age.
  Arms: IPV at 14 and 22 weeks of age, RotaTeq
Biological: IPV at 14 and fIPV at 22 weeks, Rotarix — Participants in this arm will receive a full dose of inactivated poliovirus vaccine (IPV) at 14 weeks of age and a fractional dose IPV (fIPV) booster at 22 weeks of age. They will also receive the rotavirus vaccine, Rotarix, at 6 and 10 weeks of age.
  Arms: IPV at 14 and fIPV at 22 weeks, Rotarix
Biological: IPV at 14 and fIPV at 22 weeks, RotaTeq — Participants in this arm will receive a full dose of inactivated poliovirus vaccine (IPV) at 14 weeks of age and a fractional dose IPV (fIPV) booster at 22 weeks of age. They will also receive the rotavirus vaccine, RotaTeq, at 6, 10, and 14 weeks of age.
  Arms: IPV at 14 and fIPV at 22 weeks, RotaTeq
Biological: IPV at 6 and fIPV at 22 weeks, Rotarix — Participants in this arm will receive a full dose of inactivated poliovirus vaccine (IPV) at 6 weeks of age and a fractional dose IPV (fIPV) booster at 22 weeks of age. They will also receive the rotavirus vaccine, Rotarix, at 6 and 10 weeks of age.
  Arms: IPV at 6 and fIPV at 22 weeks, Rotarix
Biological: IPV at 6 and fIPV at 22 weeks, RotaTeq — Participants in this arm will receive a full dose of inactivated poliovirus vaccine (IPV) at 6 weeks of age and a fractional dose IPV (fIPV) booster at 22 weeks of age. They will also receive the rotavirus vaccine, RotaTeq, at 6, 10, and 14 weeks of age.
  Arms: IPV at 6 and fIPV at 22 weeks, RotaTeq
Biological: fIPV at 6-14-22 weeks of age, Rotarix — Participants in this arm will receive a fractional doses of inactivated poliovirus vaccine (fIPV) at 6 and 14 weeks of age and a fIPV booster at 22 weeks of age. They will also receive the rotavirus vaccine, Rotarix, at 6 and 10 weeks of age.
  Arms: fIPV at 6-14-22 weeks of age, Rotarix
Biological: fIPV at 6-14-22 weeks of age, RotaTeq — Participants in this arm will receive a fractional doses of inactivated poliovirus vaccine (fIPV) at 6 and 14 weeks of age and a fIPV booster at 22 weeks of age. They will also receive the rotavirus vaccine, RotaTeq, at 6, 10, and 14 weeks of age.
  Arms: fIPV at 6-14-22 weeks of age, RotaTeq

SUMMARY:
This is an open-label phase IV, randomized controlled trial of inactivated poliovirus vaccine (IPV) and rotavirus vaccines. This trial will assess immunogenicity of a booster dose of fractional IPV (fIPV) in comparison with a full dose of IPV when given after varying IPV and fIPV schedules. Differences in immunogenicity of the varying schedules of IPV and fIPV will also be examined. Concomitantly, immunogenicity to two different rotavirus vaccines will be evaluated.

DETAILED DESCRIPTION:
With the switch from trivalent to bivalent oral poliovirus vaccine (OPV) in 2016, the Global Polio Eradication Initiative (GPEI) is recommending inactivated poliovirus vaccine (IPV) use as one of the potential strategies to respond to outbreaks of type 2 wild type and/or circulating vaccine-derived polioviruses. However, the current global inactivated poliovirus vaccine (IPV; 0.5 mL, full-dose) supply shortage dramatically limits the number of doses available for an effective outbreak response. Therefore, GPEI has proposed use of intradermal administration of a booster of fractional IPV (fIPV; 0.1 mL, one-fifth the full-dose) as a dose-sparing strategy to increase the number of children vaccinated and stretch IPV supplies. No study has compared immunogenicity of a fIPV booster in children previously vaccinated with a single IPV. Furthermore, the IPV shortage has led to reconsideration of fIPV use in routine immunization programs. Previous studies found that in one and two dose head-to-head comparisons, fIPV induced a lower proportion of seroconversion and antibody responses than IPV. However, recent studies of seroconversion and priming suggest two fIPV given at least eight weeks apart may be more immunogenic than one IPV. Because of these findings and the global IPV shortage, the most recent WHO position paper suggests that countries consider administering two fIPV at 6 and 14 weeks of age as an alternative to one IPV after the OPV2 cessation in April 2016. However, no trial has conducted a direct comparison of the immunogenicity of IPV at 14 weeks of age with that of fIPV at 6 and 14 weeks of age.

The immunogenicity of rotavirus (RV) vaccines will also be assessed when given concomitantly with IPV/fIPV. Currently, WHO recommends either of two licensed, live attenuated oral rotavirus vaccines for all children worldwide: the pentavalent RotaTeq (RV5) and monovalent Rotarix (RV1). Many lower income countries where IPV is being introduced are also poised to introduce rotavirus vaccine in the coming years. The first dose of OPV interferes with RV vaccines and RV vaccines may be more immunogenic when delivered with IPV compared with OPV. The proposed study presents an opportunity to compare the two and three dose responses of RV1 and RV5 when delivered with IPV compared with previous studies in Bangladesh when co-administered with OPV.

In addition, recent studies have suggested that host genetic factors (i.e., Secretor status and Lewis and salivary ABO blood group phenotype) mediate susceptibility to rotavirus infection. More precisely, non-secretors (i.e., children lacking a functional fucosyl transferse-2 [FUT2] gene) have substantially reduced risk of rotavirus infection of certain genotypes. Furthermore, certain rotavirus genotypes infected mainly Lewis negative children, independent of secretor status. In addition, blood group antigen status has been proposed to be associated with infection (or lack of infection) by particular rotavirus genotypes. The proposed trial will assess whether Secretor status, Lewis and salivary ABO blood group phenotype are also associated with vaccine response.

ELIGIBILITY:
Inclusion Criteria:

* Infants 6 weeks of age (range: 42-48 days).
* Parents that consent for participation in the full length of the study.
* Parents that are able to understand and comply with planned study procedures.

Exclusion Criteria:

* Parents and infants who are unable to participate in the full length of the study.
* A diagnosis or suspicion of immunodeficiency disorder either in the infant or in an immediate family member.
* A diagnosis or suspicion of bleeding disorder that would contraindicate parenteral administration of IPV or collection of blood by venipuncture.
* Acute diarrhea, infection or illness at the time of enrollment (6 weeks of age) that would require infant's admission to a hospital.
* Acute vomiting and intolerance to liquids within 24 hours before the enrollment visit (6 weeks of age).
* Evidence of a chronic medical condition identified by a study medical officer during physical exam.
* Receipt of any polio vaccine (OPV or IPV) before enrollment based upon documentation or parental recall.
* Receipt of any rotavirus vaccine (RV1 or RV5) before enrollment based upon documentation or parental recall.
* Known allergy/sensitivity or reaction to polio or rotavirus vaccine, or contents of polio or rotavirus vaccine.
* Infants from multiple births. Infants from multiple births will be excluded because the infant(s) who is/are not enrolled would likely receive OPV through routine immunization and transmit vaccine poliovirus to the enrolled infant.
* Infants from premature births (<37 weeks of gestation).
* History of intussusception, intestinal malformations, or abdominal surgery.

Ages: 6 Weeks to 6 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1144 (Actual)
Dates: Start 2016-09; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Immune response (yes/no) as measured by antibody titers to poliovirus types 1, 2, and 3 after vaccination with study vaccines. | Measured at 26 weeks of age.
  Immune response will be defined as either a four-fold increase in titer or a seronegative participant (<1:8 titers) who becomes seropositive (≥1:8) between designated time points. For selected objectives, baseline maternal antibody titer will be determined at 6 weeks of age and the estimated maternal antibody level at each blood collection will be calculated assuming an exponential decline with a half-life of 28 days.
Immune response (yes/no) as measured by antibody titers to poliovirus types 1, 2, and 3 after vaccination with study vaccines (priming). | Measured at 23 weeks of age.
  Priming is defined as the absence of type-specific immune response at 22 weeks with evidence of type-specific seroconversion at 23 weeks. That is, seronegative participants at 22 weeks (<1:8 titers) who become seropositive at 23 weeks (≥1:8) or a four-fold rise in type-specific antibody titers at 23 weeks compared to 22 weeks.
Immune response (yes/no) as measured by antibody titers to poliovirus types 1, 2, and 3 after vaccination with study vaccines. | Measured at 22 weeks of age.
  Immune response will be defined as either a four-fold increase in titer or a seronegative participant (<1:8 titers) who becomes seropositive (≥1:8) between designated time points. Baseline maternal antibody titer will be determined at 6 weeks of age and the estimated maternal antibody level at each blood collection will be calculated assuming an exponential decline with a half-life of 28 days.

SECONDARY OUTCOMES:
Median antibody titers at 26 weeks to poliovirus types 1, 2, and 3 | Measured at 26 weeks of age
  Median antibody titers to poliovirus types 1, 2, and 3 after vaccination with study vaccines.
Median antibody titers at 23 weeks to poliovirus types 1, 2, and 3 | Measured at 23 weeks of age
  Median antibody titers to poliovirus types 1, 2, and 3 after vaccination with study vaccines.
Median antibody titers at 22 weeks to poliovirus types 1, 2, and 3 | Measured at 22 weeks of age
  Median antibody titers to poliovirus types 1, 2, and 3 after vaccination with study vaccines.
Percentage of children achieving rotavirus IgA seroconversion | Change after completion of study vaccine series in comparison with 6 weeks of age.
  Seropositive defined as anti-Rotavirus IgA titer ≥40. Seroconversion defined as a titer ≥40 if anti-rotavirus IgA negative at 6 weeks of age (baseline) or ≥4-fold rise in titer if anti-rotavirus IgA positive at baseline, upon completion of vaccine series
Rotavirus IgA geometric mean titers | Change after completion of study vaccine series in comparison with 6 weeks of age.
Rotavirus IgA seroconversion and geometric mean titers by Secretor status, Lewis and salivary ABO blood group phenotype | Change after completion of study vaccine series in comparison with 6 weeks of age.
  Seropositive defined as anti-Rotavirus IgA titer ≥40. Seroconversion defined as a titer ≥40 if anti-rotavirus IgA negative at 6 weeks of age (baseline) or ≥4-fold rise in titer if anti-rotavirus IgA positive at baseline, upon completion of vaccine series

CONTACTS AND LOCATIONS:
Locations (1):
- International Center for Diarrhoeal Disease Research, Bangladesh, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data will not be shared beyond use by co-investigators.

REFERENCES:
- [Derived] Velasquez-Portocarrero DE, Wang X, Cortese MM, Snider CJ, Anand A, Costantini VP, Yunus M, Aziz AB, Haque W, Parashar U, Sisay Z, Soeters HM, Hyde TB, Jiang B, Zaman K. Head-to-head comparison of the immunogenicity of RotaTeq and Rotarix rotavirus vaccines and factors associated with seroresponse in infants in Bangladesh: a randomised, controlled, open-label, parallel, phase 4 trial. Lancet Infect Dis. 2022 Nov;22(11):1606-1616. doi: 10.1016/S1473-3099(22)00368-1. Epub 2022 Aug 9. PMID 35961362
- [Derived] Snider CJ, Zaman K, Estivariz CF, Yunus M, Weldon WC, Wannemuehler KA, Oberste MS, Pallansch MA, Wassilak SG, Bari TIA, Anand A. Immunogenicity of full and fractional dose of inactivated poliovirus vaccine for use in routine immunisation and outbreak response: an open-label, randomised controlled trial. Lancet. 2019 Jun 29;393(10191):2624-2634. doi: 10.1016/S0140-6736(19)30503-3. Epub 2019 May 16. PMID 31104832